CLINICAL TRIAL: NCT03970057
Title: Internet-based Cognitive Behavioural Therapy (MoodUP) in Improving Psychological Outcomes Among Perinatal Women: A Prospective Randomised Double-blind Parallel-group Trial
Brief Title: MoodUP in Improving Psychological Outcomes Among Perinatal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Collaborators: Ministry of Education, Singapore (Other Government)
Responsible Party: Principal Investigator, Lau Ying, Assistant Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NUHSRO/2017/054/T1
Record Dates: First submitted 2019-05-29; First posted 2019-05-31 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Anxiety; Pregnancy Related; Perinatal Depression; Prenatal Stress; Sleep Disturbance
Keywords: Psychological outcomes; Internet-based cognitive behavioural therapy; Perinatal women
MeSH Terms: conditions — Anxiety Disorders; Parasomnias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A randomisation algorithm on the HappyMUM website automatically assigned women to either the intervention (MoodUP) group or the control (HealthyMum) group in a 1:1 allocation ratio. A computer-generated message notified women of their group assignment. We aimed to blind women to use the active nature of the control condition. Due to the computer-based randomisation, the researchers and research assistants were unaware of the group assignment before allocation and remained blinded to the participants' group allocation throughout the trial, which ensured allocation concealment. We also blinded the group assignment to data collectors and analysts.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MoodUP (Experimental): It consisted of six weekly online sessions, homework, and forums. It covered six topics, namely managing mood, psychoeducation, cognitive restructuring, behavioural activation, lifestyle modification, and problem-solving. Each session began with an autoplay video that introduced the session goal and included video and case vignettes, short quizzes, take-home messages, and homework. We also provided an online forum for peer support and regularly monitored it.
  Interventions: Behavioral: Internet-based Cognitive Behavioural Therapy
- HealthyMUM (Placebo Comparator): It consisted of six weekly online sessions. Each session provided information on essential antenatal care using text and photos. The sessions covered topics such as parenthood, diet, exercise, breastfeeding, rest and sleep, and common problems in pregnancy.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Internet-based Cognitive Behavioural Therapy — MoodUP is an iCBT intervention that is tailored to perinatal women. The core content is presented via different types of devices, such as smartphones, tablets, laptops, or desktops, connected to the internet. The program is designed as an integration of online sessions, self-monitoring, homework, peer support, and therapist support.
  MoodUP consists of six online sessions focused on CBT skills for improving stress, anxiety, and depressive symptoms among at-risk antenatal women; each session takes between 30 and 40 minutes to complete. The content of the sessions will be as follows: Session 1: Managing mood, Session 2: Psychoeducation, Session 3: Cognitive restructuring, Session 4: Behavioural activation, Session5: Lifestyle modification, Session 6: Problem-solving.
  Other Names: MoodUP
  Arms: MoodUP
Other: Usual Care — Participants will receive a series of six, weekly online sessions comprising general antenatal education. The content of the sessions will be as follows: Session 1: Parenthood; Session 2: Diet; Session 3: Exercise; Session 4: Breastfeeding; Session 5: Rest and sleep and Session 6: Common pregnancy problems.
  Other Names: HealthyMUM
  Arms: HealthyMUM

SUMMARY:
Dramatic physiological, psychological, and social changes during the antenatal period may significantly affect a woman's psychosocial and physical conditions, thereby resulting in stress, anxiety, and depressive symptoms. Cognitive behavior therapy (CBT) is a well-established effective psychotherapy to modify thoughts, beliefs, and perceptions, as well as change the behavioral patterns under numerous conditions. However, at-risk women that need access to CBT are challenged by many issues, such as insufficient therapists, stigmatization, long waiting times, and high costs. Preventive strategies may offer a more acceptable means of addressing the problem. Internet-based CBT can help overcome some barriers to improve psychological well-being by providing a timely and efficacious intervention that is customizable, cost-effective, and flexible in terms of time and geography.

Hypotheses Compared with the control group,

1. Women who completed an internet-based CBT (MoodUP) will have significantly lower scores for stress, anxiety, and depressive symptoms immediately post-intervention and at 12 weeks post-intervention;
2. Women who completed MoodUP will reduce the frequency of negative automatic thoughts, achieve a better sleep quality, life satisfaction, and mental health immediately post-intervention and at 12 weeks post-intervention;
3. Women who completed MoodUP will have better client satisfaction.

Approach A two-stage research design will be used for 3 years. Stage I will consist of the development and validation of MoodUP based on theoretical and empirical rationales. The development of MoodUP will be guided by a combination of the basic principles from behavioral and cognitive psychology. Essential components, teaching strategies, and technical elements of MoodUP will be established according to literature review and a meta-analysis by the principal investigator and her team. Ethical and quality standards will be assessed using the Health on the Net code of conduct and the Health-Related Website Evaluation Form, respectively.

Stage II will be used to evaluate the efficacy of MoodUP among 143 antenatal women using a randomized controlled trial, two-armed parallel group pretest, and repeated post-test following the Consolidated Standards of Report Trials guidelines for an internet-based intervention. Primary outcomes will be the presence and severity of antenatal stress, anxiety, and depressive symptoms using the 21-item Depression Anxiety Stress Scale. Secondary outcomes will be automatic thoughts, sleep disturbance, life satisfaction, mental well-being, and client satisfaction, as determined by the 30-item Automatic Thoughts Questionnaires, four-item Sleep Disturbance subscale of the Medical Outcomes Study Sleep Scale, the five-item Satisfaction with Life Scale, the WHO five-item Well-Being Index, and the seven-item Client Satisfaction Questionnaire, respectively. Multivariate analysis of variance with repeated measures will be used to compare the mean difference of scores in the three-time points through Wilks's lambda test. The data will be analyzed according to the intention-to-treat principle with baseline values imputed for missing follow-up data.

ELIGIBILITY:
Inclusion Criteria:

* < 18 weeks of gestation (the upper limit of < 18 weeks allows time to complete six sessions and follow-up questionnaires prior to delivery)
* 21 years of age or older
* ability to speak and read English
* plan to deliver baby in Singapore
* can access the internet.

Exclusion Criteria:

* severe psychiatric illness
* severe medical complications
* severe obstetric complications
* fetal abnormality.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Enrollment: 368 (Actual)
Dates: Start 2021-06-04 (Actual); Primary Completion 2023-04-11 (Actual); Study Completion 2024-06-27 (Actual)

PRIMARY OUTCOMES:
Antenatal Stress | 2 years
  The DASS-21 is used to rate the frequency and severity of experiencing negative emotions over the previous week (P. F. Lovibond & S. H. Lovibond, 1995).
  Each of the three DASS-21 scales contains 7 item, divided into sub-scales of stress, anxiety and depressive symptoms (S. H. Lovibond & P. F. Lovibond, 1995).
  Frequency/severity ratings are made on a series of four-point scales from 0 (did not apply to me at all) to 3 (applied to me very much or most of the time).
  Scores of each sub-scales will be multiplied by 2 to calculate the final score. The total score ranges of each sub-scales from 0 to 42, and a high score on each sub-scale indicates more stress, anxiety and depression.
Antenatal Anxiety | 2 years
  The DASS-21 is used to rate the frequency and severity of experiencing negative emotions over the previous week (P. F. Lovibond & S. H. Lovibond, 1995).
  Each of the three DASS-21 scales contains 7 item, divided into sub-scales of stress, anxiety and depressive symptoms (S. H. Lovibond & P. F. Lovibond, 1995).
  Frequency/severity ratings are made on a series of four-point scales from 0 (did not apply to me at all) to 3 (applied to me very much or most of the time).
  Scores of each sub-scales will be multiplied by 2 to calculate the final score. The total score ranges of each sub-scales from 0 to 42, and a high score on each sub-scale indicates more stress, anxiety and depression.
Antenatal Depressive Symptoms | 2 years
  The DASS-21 is used to rate the frequency and severity of experiencing negative emotions over the previous week (P. F. Lovibond & S. H. Lovibond, 1995).
  Each of the three DASS-21 scales contains 7 item, divided into sub-scales of stress, anxiety and depressive symptoms (S. H. Lovibond & P. F. Lovibond, 1995).
  Frequency/severity ratings are made on a series of four-point scales from 0 (did not apply to me at all) to 3 (applied to me very much or most of the time).
  Scores of each sub-scales will be multiplied by 2 to calculate the final score. The total score ranges of each sub-scales from 0 to 42, and a high score on each sub-scale indicates more stress, anxiety and depression.

SECONDARY OUTCOMES:
30-item Automatic Thoughts | 2 years
  Measured through Automatic Thoughts Questionnaire. The Automatic Thought Questionnaire (ATQ) is used to measure the occurrence of negative thoughts and related cognitive processes (Hollon & Kendall, 1980).
  It consisted of 30 statements reflecting negative cognition (Hollon & Kendall, 1980). Respondents are asked to rate the frequency at which each self-statement or a similar self-statement occurred over the course of the past week.
  The responses are provided on a 5-point scale from 1 (not at all) to 5 (all the time) in order to determine the severity of symptoms. The total score ranges from 30 to 150. A high scores represents more frequent negative thoughts and cognition (Hollon & Kendall, 1980).
5-item Life satisfaction | 2 years
  Measured through The Satisfaction with Life Scale (SWLS) (Diener, Emmons, Larsen, & Griffin, 1985).
  The five-item Satisfaction with Life Scale (SWLS) is used to assess life satisfaction of the women.
  Women will rate each item on a seven-point Likert scale from 1 (strongly disagree) to 7 (strongly agree). The total score ranges from 5 to 35, and a high score on SWLS indicates high life satisfaction.
Four-item Sleep Disturbance subscale | 2 years
  Measure through Medical Outcomes Study Sleep Scale (MOSSS). The four-item sleep disturbance sub-scale of the Medical Outcomes Study Sleep Scale (Hays et al., 2005) is used to assess how well women sleep without tapping into other sleep-related medical conditions.
  Three items related to sleep disturbance are rated on a six-point Likert scale, from 1 (less than 15 minutes) to 6 (none of the time), and one item related to the time needed to fall asleep is assessed on a five-point Likert scale, from 1 (less than 15 minutes) to 5 (more than 60 minutes). Scores are converted to an index that ranged from 0 to 100, with high scores indicating a high level of sleep disturbance.
5-item Mental well-being | 2 years
  Measured through the WHO Well-Being Index (WHOWBI) (Bech, 2012; World Health Organization, 1998).
  The WHO five-item Well-Being Index is used to measure overall mental well-being. Each item is rated on a six-point Likert scale from 0 (at no time) to 5 (all of the time). The total score ranges from 0 to 25, and a high score represents better well-being.
7-item Client satisfaction | 2 years
  Measured through a self-developed questionnaire to evaluate the clients' satisfaction of website.
  Client Satisfaction Questionnaire (CSQ) is developed by our research team. Each item is rated on a four-point Likert scale from 1 to 4, and response options differed for the various items. The total score ranges from 7 to 28, and a high score represents better client satisfaction. In addition, we have four open questions to obtain suggestions for improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Lau, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Cherry, Singapore, Singapore

REFERENCES:
- [Background] Olthuis JV, Watt MC, Bailey K, Hayden JA, Stewart SH. Therapist-supported Internet cognitive behavioural therapy for anxiety disorders in adults. Cochrane Database Syst Rev. 2015 Mar 5;(3):CD011565. doi: 10.1002/14651858.CD011565. PMID 25742186
- [Background] Agius A, Xuereb RB, Carrick-Sen D, Sultana R, Rankin J. The co-existence of depression, anxiety and post-traumatic stress symptoms in the perinatal period: A systematic review. Midwifery. 2016 May;36:70-9. doi: 10.1016/j.midw.2016.02.013. Epub 2016 Mar 4. PMID 27106946
- [Background] Beck AT, Haigh EA. Advances in cognitive theory and therapy: the generic cognitive model. Annu Rev Clin Psychol. 2014;10:1-24. doi: 10.1146/annurev-clinpsy-032813-153734. Epub 2014 Jan 2. PMID 24387236
- [Background] Lau Y, Htun TP, Wong SN, Tam WSW, Klainin-Yobas P. Therapist-Supported Internet-Based Cognitive Behavior Therapy for Stress, Anxiety, and Depressive Symptoms Among Postpartum Women: A Systematic Review and Meta-Analysis. J Med Internet Res. 2017 Apr 28;19(4):e138. doi: 10.2196/jmir.6712. PMID 28455276
- [Background] Webb TL, Joseph J, Yardley L, Michie S. Using the internet to promote health behavior change: a systematic review and meta-analysis of the impact of theoretical basis, use of behavior change techniques, and mode of delivery on efficacy. J Med Internet Res. 2010 Feb 17;12(1):e4. doi: 10.2196/jmir.1376. PMID 20164043
- [Background] Hope DA, Burns JA, Hayes SA, Herbert JD, Warner MD. Automatic Thoughts and Cognitive Restructuring in Cognitive Behavioral Group Therapy for Social Anxiety Disorder. Cognitive Therapy and Research. 2010;34(1):1-12.
- [Background] Faulconbridge LF, Wadden TA, Thomas JG, Jones-Corneille LR, Sarwer DB, Fabricatore AN. Changes in depression and quality of life in obese individuals with binge eating disorder: bariatric surgery versus lifestyle modification. Surg Obes Relat Dis. 2013 Sep-Oct;9(5):790-6. doi: 10.1016/j.soard.2012.10.010. Epub 2012 Nov 14. PMID 23260806
- [Background] Ebert DD, Lehr D, Boss L, Riper H, Cuijpers P, Andersson G, Thiart H, Heber E, Berking M. Efficacy of an internet-based problem-solving training for teachers: results of a randomized controlled trial. Scand J Work Environ Health. 2014 Nov;40(6):582-96. doi: 10.5271/sjweh.3449. Epub 2014 Aug 13. PMID 25121986
- [Background] Eysenbach G. CONSORT-EHEALTH: implementation of a checklist for authors and editors to improve reporting of web-based and mobile randomized controlled trials. Stud Health Technol Inform. 2013;192:657-61. PMID 23920638
- [Background] Lovibond, S. H., & Lovibond, P. F. (1995). Manual for the Depression Anxiety Stress Scales (Second ed.). Sydney: Psychology Foundation of Australia.
- [Background] Hollon, S. D., & Kendall, P. C. (1980). Cognitive self-statements in depression: Development of an automatic thoughts questionnaire. Cognitive Therapy and Research, 4(4), 383-395. doi:10.1007/BF01178214
- [Background] Hays RD, Martin SA, Sesti AM, Spritzer KL. Psychometric properties of the Medical Outcomes Study Sleep measure. Sleep Med. 2005 Jan;6(1):41-4. doi: 10.1016/j.sleep.2004.07.006. Epub 2004 Nov 11. PMID 15680294
- [Background] Diener E, Emmons RA, Larsen RJ, Griffin S. The Satisfaction With Life Scale. J Pers Assess. 1985 Feb;49(1):71-5. doi: 10.1207/s15327752jpa4901_13. PMID 16367493
- [Background] World Health Organization. (1998). Regional Office for Europe: Wellbeing Measures in Primary Health Care: the Depcare Project. Paper presented at the Report on a WHO Meeting.
- [Background] Bech, P. (2012). Clinical Psychometrics. Oxford: Wiley-Blackwell.